CLINICAL TRIAL: NCT03384641
Title: An Open-Label Study to Evaluate the Efficacy and Safety of TMC207 in Subjects With Multibacillary Leprosy
Brief Title: A Study to Evaluate the Efficacy and Safety of Bedaquiline (TMC207) in Participants With Multibacillary Leprosy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108416; TMC207LEP2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Leprosy, Multibacillary
MeSH Terms: conditions — Leprosy, Multibacillary | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bedaquiline (Experimental): Participants will receive bedaquiline 200 (milligram) mg (2*100 mg tablets) once daily for 2 weeks followed by 100 mg tablet three times a week (tiw) for 6 weeks with at least 48 hours between doses.
  Interventions: Drug: Bedaquiline 200 mg

INTERVENTIONS:
Drug: Bedaquiline 200 mg — Participants will receive bedaquiline 200 mg (2*100 mg tablets) once daily for 2 weeks followed by 100 mg tablet tiw for 6 weeks with at least 48 hours between doses.
  Other Names: TMC207

SUMMARY:
The purpose of this study is to assess the efficacy of an 8-week bedaquiline monotherapy regimen in participants with treatment-naive, multibacillary (MB) leprosy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has: a) multibacillary (MB) leprosy, defined as 6 or more skin lesions or extensive confluent lesions or diffuse skin involvement, and is either borderline lepromatous or polar lepromatous, as determined using Ridley and Jopling classification system; and b) has a bacteriological index of >=4+ from the lesion biopsy obtained at screening, and a bacteriological index of >= 1+ from each of 4 slit skin smear assessments taken at screening
* Otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and initialed by the investigator
* Otherwise healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, including liver enzymes, other specific tests, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* a man must agree not to donate sperm throughout treatment with TMC207 and for 3 months after treatment is stopped
* Willing and able to adhere to the prohibitions, restrictions, and long-term follow up requirements specified in this protocol
* If a woman is of childbearing potential, must be practising a highly effective method of birth control (failure rate of <1% per year when used consistently and correctly) before entry, and must also agree to use a barrier contraceptive method (that is, male or female condom, diaphragm or cervical cap) plus spermicide. participant must also agree to continue to use a highly effective method of contraception plus a barrier method throughout treatment with TMC207 and until 6 months after treatment is stopped

Exclusion Criteria:

* Has experienced or is experiencing a lepra reaction requiring treatment with a prohibited therapy
* Has a contraindication limiting the implementation of a medically accepted MB leprosy regimen
* a) Has ever received pharmacotherapy for leprosy; b) has ever been treated with a drug that is a component of the primary World Health Organization (WHO) regimen for the treatment of MB leprosy (example, dapsone, rifampicin, clofazimine). Short-term (<=2 weeks) pharmacotherapy with any antibiotic that could be used as a second line treatment for leprosy (eg, of the macrolide, quinolone, or tetracycline class) is acceptable as long as the last administration occurred >=4 weeks before first dose of study drug (TMC207)
* Has a concomitant infection that requires an additional systemic antimicrobial agent
* Has tuberculosis (TB), as determined by medical history and chest x-ray
* Is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Odds of Mycobacterium leprae (M. leprae) Growth in Mouse Footpads Following 8 Weeks of Treatment with Bedaquiline | Baseline up to Week 8
  Change from baseline in the odds of M. leprae growth in mouse footpads will be evaluated. M. leprae bacilli will be inoculated in footpads of mice, according to the method of Shepard. M. leprae growth will be determined by technologists trained and experienced in mouse footpad procedures, at 1 year after infection (or at mouse death or humane endpoint, if it occurs greater than or equal to [>=] 6 months after footpad inoculation). The number of footpads with positive growth (>=10^5 M. leprae) will be counted and used to determine the odds of bacterial growth.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 124 Weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with AEs by Severity | Up to 124 Weeks
  Severity of adverse events will be graded by using division of microbiology and infectious diseases (DMID) adult toxicity scale to estimate grade of severity. Severity scale ranges from Grade 1 (Mild) to Grade 4 (Life-threatening). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, and Grade 4= Life-threatening.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Brazil (2):
  - Instituto Lauro de Souza Lima, Bauru
  - Fundacao Hospitalar de Dermatologia Tropical e Venereologia Alfredo da Matta - FUHAM, Manaus

REFERENCES:
- [Derived] Barreto J, Sammarco Rosa P, Adams L, Aguilar Z, Bakare N, Chaplan SR, Akli RD, Ernault E, Kulke S, Lounis N, Millington D, Palmer JA, Remmerie B, Wang M, Young S, Truman R, Rebello PFB. Bedaquiline Monotherapy for Multibacillary Leprosy. N Engl J Med. 2024 Dec 12;391(23):2212-2218. doi: 10.1056/NEJMoa2312928. PMID 39665652